CLINICAL TRIAL: NCT03541863
Title: What Comes After Fulvestrant? A Real World Multicenter Retrospective Study-Treatment After Progression of Fulvestrant Among Metastatic Breast Cancer Patients in China
Brief Title: Treatment After Progression of Fulvestrant Among Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-1
Record Dates: First submitted 2018-05-06; First posted 2018-05-31 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Fulvestrant; Progression; Endocrine sensitivity
MeSH Terms: conditions — Breast Neoplasms; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endocrine therapy: use endocrine therapy (ET) after Fulvestrant, include but not limited to: tamoxifen, anastrozole, letrozole, exemestane, exemestane + everolimus
- Chemotherapy: use Chemotherapy (CT) after Fulvestrant, include but not limited to: capecitabine, docetaxel-based, vinorelbine, paclitaxel-based

SUMMARY:
What Comes After Fulvestrant? A Real World Multicenter Retrospective Study-Treatment After Progression of Fulvestrant Among Metastatic Breast Cancer Patients in China.

DETAILED DESCRIPTION:
There is no evidence of treatment after progression of Ful. We retrospectively evaluated HR+, HER2- MBC patients failed on Ful 500mg as first line or second line therapy from 2014 to 2017 in 6 institutions. Treatment pattern, PFS, OS and safety were analyzed to figure out the situation and efficacy of treatment after Fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were treated with Fulvestrant between June 2014 to June 2017 as first line or second line therapy
* Patients received subsequent treatment after progressing on Fulvestrant for at least one cycle (>1 month)
* Complete medical history was available

Exclusion Criteria:

* Subsequent treatment was not standard therapy (cannot be classified into endocrine therapy/ chemotherapy)
* Medical history was incomplete

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
OS | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall survival
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 weeks

OTHER OUTCOMES:
Fulvestrant sensitivity | 6 weeks
  Time cutoff of Fulvestrant PFS related to next line ET or CT efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided